CLINICAL TRIAL: NCT01138956
Title: Study for Evaluation of the Immune Response of Visceral Leishmaniasis Patients Treated With Antimonial Pentavalent Associated to N-Acetylcysteine
Brief Title: Immune Response of Visceral Leishmaniasis PatientsTreated With Antimonial Plus N-Acetylcysteine
Acronym: VLNAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Roque Pacheco de Almeida, Universidade Federal de Sergipe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VLNAC
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Visceral Leishmaniasis; Immune Response; Treatment
Keywords: Visceral leishmaniasis; N-acetylcysteine; Antimony; Immune response
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Pentavalent antimonial, 20mg/kg/day, 28 days, IV, plus N-acetylcysteine (NAC), effervescent tablets of 600mg, tid, po.
  Interventions: Drug: N-acetylcysteine
- Group 2 (Active Comparator): Pentavalent antimonial, 20mg/kg/day, 28 days
  Interventions: Drug: Pentavalent antimonial

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine (NAC), effervescent tablets of 600mg, tid, po, 28 days
  Arms: Group 1
Drug: Pentavalent antimonial — Pentavalent antimonial, 20mg/kg/day, 28 days, IV
  Arms: Group 2

SUMMARY:
This study is designed to evaluate the immune and therapeutic responses of visceral leishmaniasis patients using N-acetylcysteine (NAC) as an adjuvant therapy to pentavalent antimony.

DETAILED DESCRIPTION:
In this study we intend to evaluate the immune and therapeutic responses of patients with visceral leishmaniasis N-acetylcysteine (NAC) as an adjuvant to standard treatment with pentavalent antimony, compared to treatment with antimonial only through a blind randomized clinical trial. Our hypothesis is that patients treated with NAC associated with pentavalent atimonial have a rapid changing of the immune responses, towards TH1, and clinical improvement when compared to patients who will use only the standard treatment

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 50 years
* Diagnosis of visceral leishmaniasis

Exclusion Criteria:

* Other acute or chronic diseases
* Use of immunosuppressive drugs
* AIDS
* History of allergy to NAC and/or pentavalent antimony

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Patient recovery from the visceral leishmaniasis after treatment | 6 months
  The cure is defined in the patient with reduced spleen and liver. Absence of fever for more than 15 days after treatment, weight gain, normalization of globulins and resolution of leukopenia and anemia.

SECONDARY OUTCOMES:
Immune response of visceral leishmaniasis patients after proposed treatment | one year
  Evaluation of the Immune response: peripheral blood mononuclear cells of patients are being obtained in ficoll-Hypaque gradient and stimulated in vitro with soluble antigen of L. chagasi to evaluate the production of cytokines (IFN-g, TNF-a. IL-10, TGF-b) before treatment, 15, 45, 180 and 360 days afterwards.

CONTACTS AND LOCATIONS:
Overall Officials: Roque P Almeida, MD, PhD, Principal Investigator — Hospital Universitário
Locations (1):
- University Hospital, Aracaju, Sergipe, Brazil